CLINICAL TRIAL: NCT03125278
Title: Patient Knowledge of Medication Indication
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A17-072
Record Dates: First submitted 2017-04-07; First posted 2017-04-24 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Medical Audit
MeSH Terms: interventions — Patient Medication Knowledge

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medication indication on the label: Patients discharged from Regions Hospital (St. Paul, MN) where we have implemented a standard process of printing the indication for all new medications on the prescription bottle.
  Interventions: Other: Medication knowledge
- No medication indication given: Patients discharged from Brigham and Women's Hospital (Boston, MA) where there is no requirement for providing information on medication indications to patients at discharge.
  Interventions: Other: Medication knowledge

INTERVENTIONS:
Other: Medication knowledge — Participants will be asked questions over the phone about their medications

SUMMARY:
This is a study to compare patient knowledge about the indications of their medications between two sites. Regions Hospital has a population of patients that receive the medication indication on the label for any new or changed medications at the time of patient discharge. Brigham Women's Health follows a standard policy of discharge medication labels including the name of the medication and instructions for use without any indication of what the medication is intended to treat. Consented patient will receive a phone call where researchers will ask about which medications they are taking and other questions about those medications.

The study population will be patients recently discharged from the hospital with 1 or more new or changed medications

ELIGIBILITY:
Inclusion Criteria

1. Hospital Medicine (HM) inpatient being discharged to home
2. Patient being discharged with ≥ 1 new or changed medications
3. English speaker

Exclusion Criteria

1. Inpatient being discharged to nursing home or TCU facility
2. Patient being discharged with no new or changed medications
3. Non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients recently discharged from the hospital with 1 or more new or changed medications.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Medication Knowledge Questionnaire | up to 5 days
  Scripted questionnaire administered on patients knowledge of their medication indications who received new, changed, or continued medications at discharge via phone call. Questions are focused on understand of relationship of the medication and what symptom or disease it is teaching.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Regions Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No